CLINICAL TRIAL: NCT04231500
Title: The Skin Microbiome in Graft Versus Host Disease Dynamics of the Skin-microbiota After Allogeneic Stem Cell Transplantation - a Predictive Marker for Graft Versus Host Disease?
Brief Title: The Skin Microbiome in Graft Versus Host Disease
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Gottfried und Julia Bangerter- Rhyner-Stiftung, Basel (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01939; sp19Mueller5
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Skin Microbiome; Graft Versus Host Disease; Graft Versus Host Disease in Skin
Keywords: allogeneic Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 4-6 mm punch biopsy will be taken from the affected skin area and a second one from a nearby unaffected part of the skin. Metagenomic sequencing of the punch biopsies will be performed. Biological material is appropriately stored for 20 years at the Division of Clinical Bacteriology/Mycology - in locked freezers in a restricted area only accessible to authorized personnel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with GVHD after allo-HSCT: Exploration of the skin-microbiota in patients with GVHD after allo-HSCT by sampling of skin swabs and a skin punch biopsy before conditioning procedure and additional skin biopsies from affected and healthy skin sites in case of GVHD
  Interventions: Diagnostic Test: Skin swabs; Diagnostic Test: Skin punch biopsies; Diagnostic Test: additional blood sampling
- patients without GVHD after allo-HSCT: Exploration of the skin-microbiota in patients without GVHD after allo-HSCT by sampling of skin swabs and a skin punch biopsy before conditioning procedure
  Interventions: Diagnostic Test: Skin swabs; Diagnostic Test: Skin punch biopsies; Diagnostic Test: additional blood sampling

INTERVENTIONS:
Diagnostic Test: Skin swabs — Pre-moistened skin swabs will be collected before the patient starts the conditioning regimens (before conditioning; start of HSCT = day 0, on the day of the transplantation an the repeated in week 4, 12, 24, 36 and 52 after allo-HSCT. The first swab serves as baseline reference (ideally taken at the earliest one week after a systemic antibiotic treatment). Swabs will be taken from the neck, back, right hip, buccal oral cavity and the genital mucosae. In patients who develop acute or chronic skin-GVHD additional swabs will be taken from affected skin at the time of diagnosis and then again according to the schedule of the non-lesioned skin swabs.
Diagnostic Test: Skin punch biopsies — During the first visit, a single skin punch biopsy will be taken to state the skin condition and microbiome before allo-HSCT. Further biopsies will only be taken in case of acute or chronic cutaneous GVHD. A 4-6 mm punch biopsy will be taken from the affected skin area and a second one from a nearby unaffected part of the skin. Before the biopsy, skin disinfection will be performed to avoid contamination with surface bacteria.
Diagnostic Test: additional blood sampling — an additional tube of blood (2.7ml) and an additional tube of serum (6ml) will be taken and frozen during visits 1, 2, 3 and 7 in the course of blood collection, in order to be able to carry out any later laboratory tests that may prove to be useful depending on the course of the study.

SUMMARY:
Based on the evidence on the impact of the intestinal microbiome on the Graft Versus Host Disease (GVHD) after allogeneic Hematopoietic Stem Cell Transplantation (allo-HSCT), it is hypothesized that the skin-microbiome may play a role in cutaneous GVHD as well. Therefore, this study aims at investigating the skin-microbiota of patients with GVHD after allo-HSCT and of patients without GVHD after allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* undergoing allo-HSCT at the University Hospital Basel

Exclusion Criteria:

* missing ability to judge
* illiteracy or lack of German, French or English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing allo-HSCT at the University Hospital Basel
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Determination of the bacterial microbiome of patients with GVHD after allo-HSCT vs. patients without GVHD after allo-HSCT | at week 4 after transplantation
  After lysis of the microbiota, the DNA is extracted for phylogenetic 16S ribosomal RNA gene sequencing (standard illumina protocol), which is considered the current gold standard to determine the bacterial microbiome
Determination of the bacterial microbiome of patients with GVHD after allo-HSCT vs. patients without GVHD after allo-HSCT | at week 12 after transplantation
  After lysis of the microbiota, the DNA is extracted for phylogenetic 16S ribosomal RNA gene sequencing (standard illumina protocol), which is considered the current gold standard to determine the bacterial microbiome
Determination of the bacterial microbiome of patients with GVHD after allo-HSCT vs. patients without GVHD after allo-HSCT | at week 24 after transplantation
  After lysis of the microbiota, the DNA is extracted for phylogenetic 16S ribosomal RNA gene sequencing (standard illumina protocol), which is considered the current gold standard to determine the bacterial microbiome
Determination of the bacterial microbiome of patients with GVHD after allo-HSCT vs. patients without GVHD after allo-HSCT | at week 36 after transplantation
  After lysis of the microbiota, the DNA is extracted for phylogenetic 16S ribosomal RNA gene sequencing (standard illumina protocol), which is considered the current gold standard to determine the bacterial microbiome
Determination of the bacterial microbiome of patients with GVHD after allo-HSCT vs. patients without GVHD after allo-HSCT | at week 52 after transplantation
  After lysis of the microbiota, the DNA is extracted for phylogenetic 16S ribosomal RNA gene sequencing (standard illumina protocol), which is considered the current gold standard to determine the bacterial microbiome
Change in skin-microbiota in lesional vs. non-lesional skin of patients with GVHD | before transplantation and at week 4, week 12, week 24, week 36 and at week 52 after transplantation
  After lysis of the microbiota, the DNA is extracted for phylogenetic 16S ribosomal RNA gene sequencing (standard illumina protocol), which is considered the current gold standard to determine the bacterial microbiome

SECONDARY OUTCOMES:
Change in inter-individual skin-microbiota in allo-HSCT patients | before transplantation and at week 4, week 12, week 24, week 36 and at week 52 after transplantation
  After lysis of the microbiota, the DNA is extracted for phylogenetic 16S ribosomal RNA gene sequencing (standard illumina protocol), which is considered the current gold standard to determine the bacterial microbiome
Change in intra-individual skin-microbiota in allo-HSCT patients | before transplantation and at week 4, week 12, week 24, week 36 and at week 52 after transplantation
  After lysis of the microbiota, the DNA is extracted for phylogenetic 16S ribosomal RNA gene sequencing (standard illumina protocol), which is considered the current gold standard to determine the bacterial microbiome
Change of the skin-microbiota in correlation with the frequency and type of posttransplant infections (e.g. episodes of bacteraemia). | before transplantation and at week 4, week 12, week 24, week 36 and at week 52 after transplantation
  After lysis of the microbiota, the DNA is extracted for phylogenetic 16S ribosomal RNA gene sequencing (standard illumina protocol), which is considered the current gold standard to determine the bacterial microbiome
Change of the composition of skin-microbiota in correlation with the severity of GVHD | before transplantation and at week 4, week 12, week 24, week 36 and at week 52 after transplantation
  After lysis of the microbiota, the DNA is extracted for phylogenetic 16S ribosomal RNA gene sequencing (standard illumina protocol), which is considered the current gold standard to determine the bacterial microbiome
Change in Dermatology Life Quality Index (DLQI) | before transplantation and at week 4, week 12, week 24, week 36 and at week 52 after transplantation
  There are 10 questions, covering the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, treatment. Each question refers to the impact of the skin disease on the patient's life over the previous week. Each question is scored from 0 to 3, giving a possible score range form 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).
Change in Worst Itch Numerical Rating Scale (WINRS) | before transplantation and at week 4, week 12, week 24, week 36 and at week 52 after transplantation
  Single-item numerical rating scale anchored at 0 and 10, on which 0 represents "no itching" and 10 represents "worst itch imaginable". The patient indicates the overall severity of itching attributable to his or her psoriatic skin condition by circling the number that best describes the worst level of itching in the past 24 hours.
Change in Eppendorf Itch Questionnaire (EIQ) | before transplantation and at week 4, week 12, week 24, week 36 and at week 52 after transplantation
  The questionnaire consists of two pages, which are filled in by the patient. Form 1 presents 80 randomized descriptors. Sensory items are grouped on the left side and more affective or emotional items of different intensity values are found on the right side. Every item is scored within the range of 0 ('not true') to 4 ('describes exactly my itch sensation'). Statistically evaluable intensities can be derived from form 1 for every item. Form 2 deals with temporary and topographic aspects. Anti-itch ('pruritofensive') measures are grouped here and itch intensity is rated on a visual analog scale.
Change in Hospital Anxiety and Depression Scale (HADS) | before transplantation and at week 4, week 12, week 24, week 36 and at week 52 after transplantation
  The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. Scores of greater than or equal to 11 on either scale indicate a definitive case.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Mueller, PD Dr. med, Principal Investigator — Department of Dermatology; University Hospital Basel
Locations (1):
- Department of Dermatology; University Hospital Basel, Basel, Switzerland